## STATISTICAL ANALYSIS PLAN

Title: The Effect of Mild Exercise While Receiving Chemotherapy on the Psychology of

the Cancer Patient

NCT Number: NCT06943638

Date: 31 July 2025

### 1. Purpose

This SAP outlines the pre-specified statistical methods for analyzing the impact of a mild exercise intervention on state anxiety levels among cancer patients undergoing chemotherapy.

### 2. Study Objectives (Statistical)

- Assess the change in STAI-Y1 anxiety scores before and after the intervention.
- Explore associations between age, gender, and anxiety score changes.

### 3. Study Variables

#### Primary Outcome:

Change in STAI-Y1 scores (post-intervention minus baseline)

#### Covariates:

Age, gender

#### 4. Statistical Methods

## Descriptive Statistics:

Summary statistics (mean, SD, median, IQR) will be calculated for all variables.

#### Inferential Tests:

- Wilcoxon signed-rank test to compare pre- and post-intervention anxiety scores (due to expected non-normal distribution).
- o Cohen's D for paired samples to assess effect size.
- Spearman's rank correlation to explore relationships between demographics and anxiety change.

# 5. Sample Size Estimation

Based on similar studies (e.g., Moraes et al., 2021), a minimum of 45 participants is estimated to provide 80% power to detect significant differences ( $\alpha$  = 0.01).

# 6. Handling of Missing Data

Any missing questionnaire responses will be evaluated. If fewer than 5% of responses are missing, listwise deletion will be used. Otherwise, imputation methods may be considered.

#### 7. Software

All analyses will be conducted using SPSS v29.